CLINICAL TRIAL: NCT01300676
Title: The Effect of Tualang Honey and Hormonal Replacement Therapy (HRT) on Safety Profiles Among Postmenopausal Women
Brief Title: The Effects of Tualang Honey on Postmenopausal Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Associate Professor Dr Nik Hazlina Nik Hussain, USM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: (USMKK/PPP/JEPeM (198.3(11)); (USMKK/PPP/JEPeM (198.3(11)) (Other: Universiti Sains Malaysia)
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2007-11

CONDITIONS: Postmenopausal Syndrome
Keywords: Tualang honey; HRT; safety profiles; cardiovascular parameters; hormonal levels; bone changes; postmenopausal women
MeSH Terms: interventions — Estradiol; Dydrogesterone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tualang Honey (Active Comparator): Group 1: Subjects receiving 20 g/day of Tualang honey. The honey used was from a single batch honey supplied by Federal Agricultural Marketing Authorities (FAMA), Malaysia, evaporated by FAMA to achieve a water content of about 20%, submitted to Sterile Gamma company at Shah Alam, Selangor for sterilization at 25 kGy and packed in 20 g sachet in collaboration with School of Pharmaceutical Sciences laboratory.
  Interventions: Drug: Tualang honey
- Group 2 (No Intervention): Group 2: Subjects receiving hormonal replacement therapy (Femoston®), also known as Femo conti 1/5 (contain 1 mg Estradiol valerate and 5 mg Dydrogesterone) supplied by Solvay Pharma Malaysia.
  Interventions: Drug: Tualang honey

INTERVENTIONS:
Drug: Tualang honey — This was a randomized, prospective, clinical study to evaluate the effect of Tualang honey in comparison with HRT. Subjects will be confined to healthy postmenopausal women who were naturally menopause for more than one year. The study period was four months. A total of 79 patients were recruited.
  Group 1: Subjects receiving 20 g/day of Tualang honey. The honey used was from a single batch honey supplied by Federal Agricultural Marketing Authorities (FAMA), Malaysia, evaporated by FAMA to achieve a water content of about 20%, submitted to Sterile Gamma company at Shah Alam, Selangor for sterilization at 25 kGy and packed in 20 g sachet in collaboration with School of Pharmaceutical Sciences laboratory.
  Group 2: Subjects receiving hormonal replacement therapy (Femoston®), also known as Femo conti 1/5 (contain 1 mg Estradiol valerate and 5 mg Dydrogesterone) supplied by Solvay Pharma Malaysia.
  Other Names: Femo conti 1/5 (contain 1 mg Estradiol valerate and 5 mg Dydrogesterone)

SUMMARY:
Despite evidence supporting the benefits of hormone replacement therapy (HRT), only 15% of postmenopausal women currently use HRT (1). The leading reasons why women refuse or discontinue HRT are fear of malignancy, side effects such as vaginal bleeding, weight gain, depressed mood, and breast tenderness, and social reasons such as regarding menopause as a natural transition, not as a disease that requires treatment. Millions of women expressed their concern on the safety of hormone replacement therapy since the data from the Women's Health Initiative (WHI) study was released, which reported an increased risk of cardiovascular disease, breast cancer, stroke and thromboembolic disease with conjugated equine estrogen plus medroxyprogesterone acetate compared with placebo (2). The study has also demonstrated that quality of life (3) and cognition (4) were no better in the HRT group than the placebo group. In view of these problems, women are increasingly turning to alternative therapies in an effort to manage their menopausal symptoms (1).

Menopause is associated with decreasing sex steroid levels. The effect of menopause on circulating androgen levels has been studied by several investigators with variable findings. The levels of testosterone and androstenedione appear to show a small but significant decrease just before or within the first 2 years after menopause, with a decrease in testosterone amounting to approximately 15% (5,6). Unlike the abrupt decrease in estradiol levels associated with menopause, circulating testosterone, DHEA, and DHEAS levels decrease more gradually, beginning in the years before menopause and continuing thereafter (6,7). As a consequence, some women may experience symptoms of androgen decrease in the period before cessation of menses. By giving Tualang Honey to these postmenopausal women, it is postulated that the symptoms of androgen deficiency or menopausal symptoms should be reduced.

The investigators have also reported that tualang honey given to ovariectomised rats, an animal model for postmenopausal states for two weeks significantly increased the free testosterone and progesterone plasma levels, but no significant effect was seen in the beta-estradiol level. There were significant increased in the thickness of vaginal epithelium and vaginal epithelial-muscular layers. Proliferation of the squamous epithelium with vacuolation of some of the squamous cells were noted in the honey treated animals implying that there were increased in mucopolysacharide content. Uterine weight, endometrial and circular muscle thickness were significantly increased in honey treated animal with cystic changes noted over the glands (8).

To date, there are no clinical studies looking at the effects of Tualang Honey on perimenopausal women. In view of the initial evidence that it is a phytoestrogen from animal studies and has androgenic properties as well, it should have a beneficial effect to these women in terms of improvement in their menopausal symptoms, changes in their endogenous hormonal profile and increase in bone mineral density.

DETAILED DESCRIPTION:
OBJECTIVES

1. To evaluate the safety profile of honey in term of haematological and biochemical profile

   * haematological function
   * liver function
   * renal function
2. To assess the changes in cardiovascular parameters

   * blood pressure
   * waist circumference
   * total cholesterol
   * high density lipoprotein
   * low density lipoprotein
   * fasting glucose
3. To assess the effects on hormonal level

   * follicular stimulating hormone (FSH)
   * luteinizing hormone (LH)
   * testosterone
   * estradiol
4. To assess the effects on bone density through bone densitometry (DEXA) scan measurement.

   Description of Methodology Study Subjects

   This is a randomized, prospective, clinical study to evaluate the effects of honey in comparison with hormone replacement therapy (HRT). Subjects will be confined to postmenopausal women. The study period will be four months, 41 subjects will be recruited for each group. A total of 82 patients will be recruited in this study. Eligible subjects consenting to participate will be randomly assigned to one of the two groups:

   GROUP 1: Subjects receiving 20 g/day of Tualang Honey GROUP 2: Subjects receiving hormonal replacement therapy (Femoston)

   Study Schedule

   About 10 ml of fasting blood samples will be collected for hormonal profiles at baseline and at the end of the study. The hormones to be assayed will be serum follicle stimulating hormone (FSH), Luteinising Hormone (LH), estradiol and total testosterone. Blood will also be taken for safety profile (haematology, liver function test and liver function test) and for cardiovascular parameters such fasting lipids and fasting blood sugar. Bone density will be check using Dual Energy X-ray Absorptiometry (DEXA) at baseline and end of the study. Subjects will be thoroughly examined by Medical Specialists who are part of the Clinical Trial Team at every 2-monthly visit.

   SAMPLE SIZE ESTIMATION

   The calculated sample size for the study is based on a standard statistical approach, often called as power calculations, which is widely used to calculate sample size in clinical trials.

   The formula is as below:

   N = p1 x (100 - p1) + p2 x (100-p2) x f (α, β)

   (p1 - p2) 2

   In our pre-clinical trial (ovariectomised rat), about 40% increase in mean testosterone level was observed among the low dose group. Assuming a similar increase of ~10% is also obtained in the placebo group, and at a power of 80%, the calculated number of subjects per group would be 29. Taken into consideration that there will be about 40% drop-out rate, each treatment group would therefore be 41 subjects.

   Actual calculation:

   Set p1 = 40; p2 = 10; α β = 7.9

   N = 40 (100-40) + 10 (100-10) x 7.9 = (40 x 60 + 10 x 90) x 7.9 (40-10)2 900

   = 29
   * 40% dropout = 29+ 12 =41 subjects per treatment arm There will be 2 groups, 41 subjects X 2 groups = Total of 82 patients need to be recruited.

   STUDY PROCEDURE Pre study screening

   Informed consent

   Healthy females, who have been considered for entry into the study, will be informed about the study and asked if they would like to participate. Subjects agreeing to participate must provide informed consent prior to any study specific assessments or procedures being informed.

   The study will be fully explained to the subject by the investigator. The investigator will provide the subject with a comprehensive explanation of the proposed treatment including , but not limited to, the nature of the therapy, alternative therapies, any known previously experienced adverse reactions, the investigational status of the tested extract and also the study aims, methods, anticipated benefits and potential hazards of the study, including any discomfort they may experience as a result of study participation. A summary of this information will also be provided to the subject in writing.

   The subject must have the opportunity to clarify with the Investigator any issues they did not understand and if necessary, ask further questions. The subject must be given adequate time to consider whether they wish to participate in the study. The subject must be informed that they are to withdraw consent at any time, without penalty or loss of benefits to which the patient is otherwise entitled.

   The investigator will obtain the subject's informed consent. The person, who obtains the informed consent, signed and dated the informed consent form. If this person is not the investigator, then the investigator must also sign and personally date the written informed consent form. A copy of the patient information sheet and the signed consent form must be provided to each subject.

   Screening procedures

   The following assessments were performed for all subjects during the screening process and recorded in the Clinical Record Form
   * Subject initials
   * Demographic details including weight and height
   * Physical examination and investigations including pelvic ultrasonography and DEXA
   * Brief medical history relating to past and current illnesses
   * Concomitant medication
   * Collect fasting blood sample for the following laboratory evaluations.

   Patient randomisation/blinding

   Subject will be randomized using Block Randomization. The assignment of Tualang Honey will be blinded to patients using ID numbers.

   Patient's withdrawal

   The investigator may cease study treatment and withdrew the subject or the subject may withdraw herself from participation in the study at any time. The reason for the withdrawal of a patient will be recorded in the CRF. Subject will be followed-up for a minimum of 30 days following the last dose of study drug.

   Possible reasons for patient withdrawal include:
   * The need to take medication, which may interfere with study measurements.
   * Patient experiences an intolerable / unacceptable adverse event
   * Patient exhibits non-compliance with the protocol
   * Patient unwilling to proceed and / or consent is withdrawn
   * Investigator withdraws patient for reasons unrelated to the study drug (e.g. undercurrent illness)

   SAFETY ASSESSMENT

   Protocol specific clinical assessment

   Screening day and end of treatment

   Demographic details will be recorded at screening. The subject's body weight, blood pressure will be measured at 2 monthly periods.

   Medical history and adverse events

   At the screening visit, a physical examination will be conducted to determine the patient's current medical conditions and past clinically significant events. This includes all events that have occurred within the last three months and any other earlier event related to the inclusion and exclusion criteria or the subject's disease. This will be recorded at the screening visit. Throughout the study period, subject will be directly questioned about the occurrence of any new signs and symptoms and any changes from baseline will be recorded as an adverse event. Diary will be given to the patient to chart the proper timing and date for ingestion of honey.

   A physical examination will be repeated at the end of the treatment and exit evaluation to assist in determining if there had been any changes to the patient's health during the study period. Physical examination details will not be recorded in the CRF, unless there are changes from the baseline that warrant recording as a new adverse event or change to an existing adverse event.

   Vital signs

   All visits

   Vital signs (supine blood pressure, pulse rate) will be recorded at every visit. Patient is supine or semi-recumbent for five minutes prior to evaluating vital signs.

   Concomitant medication

   Concomitant medication included all co-administered drugs and treatment such as analgesics, tonics, herbals or traditional medicines and vitamin and/or mineral supplements. All concomitant medication taken within 7 days prior to commencement of study drug administration and for the duration of the study will be recorded in the CRF, including indication, dose, frequency, date and route administered.

   SAFETY REPORTING

   Adverse event definition

   An adverse event (AE) is defined as any untoward medical occurrence (including clinically significant laboratory findings) in a patient or clinical investigation subject administered a pharmaceutical drug, and which did not necessarily have a causal relationship to the treatment. Adverse event may include:
   * The significant worsening of the disease or symptoms of the disease under investigation following administration of the drug
   * Any undercurrent illness with an onset after administration of the drug
   * Exacerbation (i.e. increase in frequency or intensity) of a pre-existing condition or event

   Serious adverse event definition

   A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose:

   Results in death
   * Is life-threatening. A ' life-threatening' adverse event refers to an event, which puts the patient at risk of death. It does not refer to an event, which hypothetically might cause death if it is more severe.
   * Requires in-patient hospitalization or prolongation of existing hospitalization. Hospitalization is defined as the patient being hospitalized overnight, or the patient's hospital stay being prolonged for at least an additional overnight stay. Hospital admissions for elective surgery, for social reasons or for normal disease management procedures that are not the result of the worsening of an underlying condition will not be considered a serious adverse event.
   * Results in persistent or significant disability/incapacity
   * Is a congenital anomaly/birth defect
   * Is a malignancy
   * Is the result of an overdose? An important medical event, which jeopardizes the patient and may require medical or surgical intervention to prevent one of the above outcomes from occurring.

   STATISTICAL ANALYSIS:

   Data will be entered, cleaned and analyzed using SPSS version 12. Means and standard deviations for numerical variables and frequency and proportion for categorical variables will be reported along with histogram or bar chart if necessary.

   For univariable analysis the independent t-test and one way ANOVA will be used to compare numerical outcome variables among the three treatment groups and chi square for categorical outcome variables.

   For mutivariable analysis, repeated measure ANOVA will be used for analysis to adjust for confounding variables. Level of significance is set at 5% and results will be presented with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 45 and less than 65 years old
* No present active medical, surgical and gynaecological problems
* Body mass index 18-35 kg / m2
* Not on hormone replacement therapy for more than 3 months
* Subject who has given written informed consent to participate in the study and understand the nature of the study
* Not illiterate

Exclusion Criteria:

* Taking any form of herbal extract in the last 3 months before study entry.
* History of drug or alcohol abuse.
* Following ovariectomy.
* History of breast or cervical carcinoma.
* Taking medication that affect bone metabolism, including glucocorticoid, anticonvulsant and methotrexate.
* Clinical relevant cardiovascular, gastrointestinal, hepatic, neurologic, endocrine, haematologic or other major systemic diseases making implementation of the protocol or other interpretation of the study result difficult.
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study.
* Evidence of uncooperative attitude, including poor compliance
* Inability to attend follow-up visit.
* Subject with any other medical condition (for example uncontrolled infection) that may, in the opinion of the Investigator, interfere with the study objective.
* Endometrial thickness more than 0.5 cm detected from pelvic ultrasonography.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
changes in haematological function | 4 months
  To evaluate the safety profile of honey in term of haematological and biochemical profile
changes in liver function | 4 months
  To evaluate the safety profile of honey in term of haematological and biochemical profile
changes in renal function | 4 months
  To evaluate the safety profile of honey in term of haematological and biochemical profile

SECONDARY OUTCOMES:
changes in cardiovascular parameters | 4 months
  To assess the changes in cardiovascular parameters
  * blood pressure
  * waist circumference
  * total cholesterol
  * high density lipoprotein
  * low density lipoprotein
  * fasting glucose
changes in hormonal level | 4 months
  * follicular stimulating hormone (FSH)
  * luteinizing hormone (LH)
  * testosterone
  * estradiol
changes in bone density | 4 months
  To assess the effects on bone density through bone densitometry (DEXA)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Unit, Hospital USM, Kubang Kerian, Kelantan, Malaysia